CLINICAL TRIAL: NCT07405125
Title: Safety of Robotic Surgery for Gastrointestinal Stromal Tumors at Special Anatomic Sites: A Multicenter, Prospective Clinical Study
Brief Title: Safety of Robotic Surgery for GISTs at Special Anatomic Sites
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JROS-002; 2025-SR-793 (Other: Jiangsu people hospital)
Record Dates: First submitted 2026-01-19; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Gastrointenstinal Stromal Tumor (GIST)
MeSH Terms: interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic group (Experimental)
  Interventions: Procedure: Robotic Surgery

INTERVENTIONS:
Procedure: Robotic Surgery — To perform robotic radical surgery with the aim of achieving R0 resection.

SUMMARY:
This study is a prospective, multicenter, single-arm, phase II clinical trial. It plans to enroll 182 patients with localized gastric gastrointestinal stromal tumors (GISTs) at special anatomic sites. Eligible patients who meet the inclusion/exclusion criteria and provide written informed consent will undergo robotic radical surgery. Postoperative treatment will be determined jointly by the clinicians and patients based on actual clinical practice.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumor (GIST) is the most common mesenchymal tumor of the digestive tract. For localized gastric GISTs, surgical resection remains the cornerstone of curative treatment, adhering to the fundamental principles of complete tumor excision (R0 resection), avoidance of rupture, and negative surgical margins. Since GIST rarely metastasizes to lymph nodes, local resection has become the standard procedure.

With advancements in minimally invasive techniques, laparoscopic and robotic surgeries are increasingly utilized in GIST management. International guidelines (NCCN, ESMO) and Asian consensus statements recommend laparoscopic surgery for small tumors (<5 cm) in favorable anatomic locations (e.g., gastric anterior wall, greater curvature), highlighting benefits such as reduced intraoperative bleeding, lower complication rates, and faster postoperative recovery. However, the applicability of minimally invasive techniques for tumors in special anatomic sites (e.g., cardia, pyloric region) remains controversial.

For instance, subcardiac GISTs, due to their proximity to the gastroesophageal junction (GEJ) and critical vascular structures, present significant surgical challenges. Traditional laparoscopic techniques may encounter limitations such as restricted operating space and difficulty in tumor exposure, while excessive resection may lead to loss of cardiac function or postoperative stenosis.

Robotic surgical systems, leveraging advantages like three-dimensional high-definition visualization, enhanced instrument flexibility, and tremor filtration, show unique potential for operations within confined anatomic spaces. Compared to conventional laparoscopy, its wristed instruments allow for more precise tumor dissection, potentially reducing injury to adjacent tissues. Stable visual control facilitates R0 resection in complex areas, making it particularly suitable for anatomically challenging regions (e.g., cardia, gastric posterior wall, duodenum). Some retrospective studies report successful preservation of cardiac and pyloric function with R0 resection using robotic surgery. For example, a single-center study involving 25 patients with gastric GISTs in challenging locations like the GEJ and lesser curvature undergoing robot-assisted partial gastrectomy reported preserved cardiac and pyloric function in all cases without tumor rupture. Small-sample studies also confirm that robotic resection for GISTs in the cardia or duodenum can precisely preserve cardiac and ampullary structures, avoiding the need for cardiectomy or pancreaticoduodenectomy.

Nevertheless, existing research primarily focuses on the overall efficacy of laparoscopic or robotic techniques, lacking systematic data on the success rate of robotic surgery specifically for gastric GISTs in special anatomic sites.

Although the safety of laparoscopic surgery for GISTs in certain special locations (e.g., gastric anterior wall, greater curvature) is supported by some retrospective studies, the potential advantages of robotic surgery in such cases-such as higher rates of function preservation and lower conversion rates to open surgery-remain unclarified. For instance, a multicenter study comparing open, laparoscopic, and robotic resections for gastric GIST found no significant differences in operative time or blood loss between the robotic and laparoscopic groups but did not specifically analyze cases involving special anatomic sites. Another study suggested that robotic surgery might facilitate more precise resection in difficult locations like the GEJ, but more specific, targeted evaluations are lacking.

Therefore, this study aims to prospectively analyze the application of robotic surgery for gastric GISTs in special anatomic sites, focusing on evaluating its safety and success rate, thereby addressing gaps in current guidelines and literature. The findings are expected to provide evidence-based support for the broader adoption of robotic surgery in these complex cases and potentially contribute to expanding the indications for minimally invasive techniques.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years, regardless of sex.
* Diagnosis of GIST located at a special anatomic site confirmed preoperatively by endoscopy/endoscopic ultrasound, CT, or MRI.
* Preoperative imaging suggests a tumor diameter between 2 cm and 5 cm.
* No prior neoadjuvant therapy (e.g., imatinib) administered.
* Expected survival period ≥ 6 months.
* Preoperative assessment indicates feasibility for robotic surgery.
* Preoperative examinations show no evidence of distant metastasis or direct invasion into adjacent organs.
* Preoperative ECOG Performance Status score of 0 or 1.
* Preoperative ASA Physical Status classification of I to III.
* The subject has read and fully understood the patient information sheet and provided written informed consent.

Exclusion Criteria:

* History of previous upper abdominal surgery (except laparoscopic cholecystectomy).
* History of previous gastrectomy, endoscopic mucosal resection (EMR), or endoscopic submucosal dissection (ESD).
* Previous administration of neoadjuvant therapy (e.g., imatinib).
* Presence of other active malignancies within the past 5 years or concurrently. (Note: Patients with cured localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, carcinoma in situ of the prostate, cervical carcinoma in situ, breast carcinoma in situ, Stage I lung cancer, or Stage I colorectal cancer, may be enrolled.)
* Requirement for concurrent surgery for other diseases.
* Emergency surgery performed due to tumor-related complications (bleeding, obstruction, or perforation).
* Arterial/venous thrombotic events within 6 months prior to screening, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis (excluding thrombosis related to prior chemotherapy venous catheters deemed resolved by the investigator), and pulmonary embolism.
* Myocardial infarction within 6 months prior to surgery, or poorly controlled arrhythmia (including QTc interval ≥450 ms for males or ≥470 ms for females, calculated using Fridericia's formula).
* Cardiac insufficiency classified as NYHA Class III-IV, or left ventricular ejection fraction (LVEF) <50% on cardiac ultrasound.
* Ventilatory dysfunction: FEV1 <50% of predicted value.
* Clinically symptomatic pleural or abdominal effusion requiring clinical intervention.
* Human Immunodeficiency Virus (HIV) infection.
* Active pulmonary tuberculosis.
* History or presence of interstitial lung disease, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, or severely impaired pulmonary function that may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* Any active infection requiring systemic anti-infective therapy within 14 days prior to surgery; except for prophylactic antibiotic therapy (e.g., for urinary tract infection or chronic obstructive pulmonary disease).
* Concurrent participation in another clinical trial involving surgical treatment.
* History of alcohol abuse, drug abuse, or substance abuse. (Note: Patients who have ceased alcohol consumption may be enrolled.)
* Patients deemed likely to be non-compliant with medical advice or medication regimens, or with incomplete data that may affect efficacy or safety assessment.
* Pregnant or lactating female patients.
* Any condition that may increase the risk associated with study participation, or other severe, acute, or chronic diseases, or any other situation that, in the investigator's judgment, makes the patient unsuitable for clinical study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2026-02-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival rate (3-year DFS) | Patients were followed for 3 years after undergoing robotic surgery.
  The proportion of patients who develop tumor recurrence among all patients who underwent surgery is calculated at the 3-year mark following the date of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University (Jiangsu Province Hospital), Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data and statistical analysis code
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD and supporting information will be available starting in January 2029 for two years.
Access Criteria: Interested investigators may request access by contacting zhqsq@qq.com via email. The information available includes detailed study protocol, primary outcome data, as well as analysis results and procedures.

REFERENCES:
- [Background] 1.Open and minimally invasive surgery for gastrointestinal stromal tumours a systematic review and network meta-analysis protocol. BMJ Open. 2022;12(2):e050414. 2.Robotic Function-Preserving Resection of Gastric Gastrointestinal Stromal Tumor. J Surg Res. 2023 Oct:290:164-170. 3.Application of Intragastric Single-Incision Laparoscopy Surgery in the Management of Gastroesophageal Junction Gastrointestinal Stromal Tumors. J Vis Exp. 2025 Jun 17:(220) 4.Robotic excision of gastric and duodenal gastrointestinal stromal tumor. Updates Surg. 2022 Aug;74(4):1483-1484. 5. Laparoscopic and robot-assisted procedures in patients with gastrointestinal stromal tumors (GIST) of stomach. Khirurgiia (Mosk). 2020:(1):5-13. 6.Robotic limited local resection of duodenal juxta-ampullary neoplasms. Int J Med Robot. 2021 Apr;17(2):e2192. 7.Robotic duodenal (D3) resection with Roux-en-Y duodenojejunostomy reconstruction for large GIST tumor Step by step with video. Surg Oncol. 2021 Mar:36:130. 8.Is minimally invasive surgery for large gastric GIST actually safe? A comparative analysis of short- and long-term outcomes. Surg Endosc. 2022 Sep;36(9):6975-6983 9.Pylorus resection versus pylorus preservation in pancreatoduodenectomy (PyloResPres) study protocol and statistical analysis plan for a German multicentre single-blind surgical registry-based randomised controlled trial. BMJ Open. 2021 Nov 29;11(11):e056191 10.Robot-assisted laparoscopic combined with endoscopic partial gastrectomy (RALE-PG) for the treatment of gastric gastrointestinal stromal tumors in challenging anatomical locations single-center experience. Front Surg. 2024 May 23:11:1391387. 11.Oncologic outcomes and survival of modern surgical approaches for gastric gastrointestinal stromal tumor (GIST). Surg Endosc. 2024 Nov;38(11):6854-6864. 12.Open versus laparoscopic versus robotic gastric gastrointestinal stromal tumour resections A multicentre cohort study. Int J Med Robot. 2021 Apr;17(2):e2198.